CLINICAL TRIAL: NCT00552240
Title: Comparison Atazanavir/Ritonavir (ATV/r) vs Nevirapine (NVP) Twice a Day (Bid) on Truvada Backbone
Brief Title: Nevirapine vs. Atazanavir Boosted With Ritonavir on a Background of Truvada in Human Immunodeficiency Virus (HIV) Infected Naive Patients (NEwArT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1512
Record Dates: First submitted 2007-09-28; First posted 2007-11-01 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Nevirapine; BID protein, human; Atazanavir Sulfate; Ritonavir

ARMS (2):
- NVP 200mg bis indie (BID) (Active Comparator): after receiving nevirapine (NVP) 200 mg quaue die (QD) for 2 weeks, pt titrated to NVP 200 mg bis in die (BID) combined with emtricitabine 200 mg QD/ tenofovir DF 300 mg QD (fixed dose combination Truvada) for 48 weeks
  Interventions: Drug: tenofovir DF 300 mg QD; Drug: emtricitabine 200 mg QD; Drug: Nevirapine 200 mg BID
- Atazanavir 300 mg QD/ritonavir 100 mg QD (Active Comparator): patients to receive atazanavir 300 mg QD boosted with ritonavir 100 mg QD combined with emtricitabine 200 mg QD/ tenofovir DF 300 mg QD (fixed dose combination Truvada) for 48 weeks
  Interventions: Drug: tenofovir DF 300 mg QD; Drug: emtricitabine 200 mg QD; Drug: Atazanavir 300 mg; Drug: Ritonavir 100 mg

INTERVENTIONS:
Drug: tenofovir DF 300 mg QD — 300 mg QD
  Arms: Atazanavir 300 mg QD/ritonavir 100 mg QD
Drug: tenofovir DF 300 mg QD — 300 mg QD
  Arms: NVP 200mg bis indie (BID)
Drug: emtricitabine 200 mg QD — 200 mg QD
  Arms: Atazanavir 300 mg QD/ritonavir 100 mg QD
Drug: emtricitabine 200 mg QD — 200 mg QD
  Arms: NVP 200mg bis indie (BID)
Drug: Nevirapine 200 mg BID — 200 mg BID
  Arms: NVP 200mg bis indie (BID)
Drug: Atazanavir 300 mg — 300 mg QD
  Arms: Atazanavir 300 mg QD/ritonavir 100 mg QD
Drug: Ritonavir 100 mg — 100 mg QD
  Arms: Atazanavir 300 mg QD/ritonavir 100 mg QD

SUMMARY:
The aim of this clinical trial is to compare the efficacy and safety of ritonavir (RTV)-boosted atazanavir with nevirapine, each on a background of emtricitabine and tenofovir disoproxil fumarate (DF).

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent in accordance with Good Clinical Practice (GCP) and local regulatory requirements prior to trial participation
2. HIV-1- infected males or females greater than or equal to 18 years of age with documented positive serology Enzyme-linked Immuno Sorbert Assay (ELISA) confirmed by Western blot
3. No prior nucleoside reverse transcriptase inhibitor (NRTI) or non-nucleoside reverse transcriptase inhibitor (NNRTI) use of more than 10 days AND
4. No prior use of other classes of antiretrovirals (ARVs) of more than 2 weeks duration
5. Males with CD4+ count less than 400 cells/mm cubed or females with CD4+ count less than 250 cells/mm cubed
6. NVP and ATV/r susceptibility on screening HIV-1 genotypic resistance assay
7. Adequate renal function defined as a calculated creatinine clearance greater than or equal to50 ml/min according to the Cockcroft-Gault formula
8. Karnofsky score greater than or equal to 70 (see Appendix 10.7)
9. Acceptable medical history, as assessed by the investigator

Exclusion criteria:

1. History of active drug or alcohol abuse within 2 years prior to study entry (at the investigators discretion)
2. Hepatic cirrhosis with stage Child-Pugh B or C hepatic impairment
3. Female patients of child-bearing potential who:

   have a positive serum pregnancy test at screening, are breast feeding, are planning to become pregnant, are not willing to use a barrier method of contraception, or are not willing to use methods of contraception other than ethinyl estradiol containing oral contraceptives
4. Laboratory parameters greater than Division of Aids (National Institute of Health, USA) (DAIDS) grade 2 (triglycerides greater than DAIDS grade 3, total cholesterol no restrictions, see Appendix 10.1)
5. Active hepatitis B or C disease, defined as HBsAg-positive or Hepatitis C Virus (HCV) RNA positive with alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ALT/AST greater than2.5x Upper Limit of Normal (ULN) (greater than DAIDS grade 1)
6. Known hypersensitivity to any ingredients in nevirapine or atazanavir
7. Patients who are receiving concomitant treatments which are not permitted, as listed in Appendix 10.6
8. Use of other investigational medications within 30 days before study entry or during the trial
9. Use of immunomodulatory drugs within 30 days before study entry or during the trial (e.g., interferon, cyclosporin, hydroxyurea, interleukin 2, chronic treatment with prednisone)
10. Patients with Progressive Multifocal Leukoencephalopathy (PML), visceral Kaposi's Sarcoma (KS), and/or any lymphoma
11. Any AIDS defining illness that is unresolved, symptomatic or not stable on treatment for at least 12 weeks at the screening visit
12. Patients who are receiving systemic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- United States (19):
  - 1100.1512.28 Boehringer Ingelheim Investigational Site, Beverly Hills, California
  - 1100.1512.20 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1100.1512.15 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1100.1512.26 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 1100.1512.17 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1100.1512.14 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1100.1512.23 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 1100.1512.29 Boehringer Ingelheim Investigational Site, Maywood, Illinois
  - 1100.1512.11 Boehringer Ingelheim Investigational Site, Neptune City, New Jersey
  - 1100.1512.25 Boehringer Ingelheim Investigational Site, Newark, New Jersey
  - 1100.1512.18 Boehringer Ingelheim Investigational Site, Somers Point, New Jersey
  - 1100.1512.22 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1100.1512.21 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1100.1512.13 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1100.1512.30 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1100.1512.19 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1100.1512.16 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1100.1512.24 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1100.1512.27 Boehringer Ingelheim Investigational Site, Annandale, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 28 Sep 2007 through 23 Mar 2009 at 18 sites throughout the US. The sites were comprised of medical centers or private practice physicians.
Pre-assignment Details: There was a 28 day screening period where a genotype report was run. If patients were resistant to any of the study medication, they were not to be randomized into the study. Patients also needed to meet all inclusion/exclusion criteria in order to be eligible. 154 patients were enrolled but 2 were not treated, leaving 152 in full analysis set.
Groups:
- Nevirapine (NVP) Plus Truvada: Nevirapine 200 mg bis in die (BID)
- Atazanavir Plus Ritonavir (ATV/r) Plus Truvada: Atazanavir 300 mg plus ritonavir 100 mg quaque die (QD)
Period: Overall Study
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Started | 75 (Number in Full Analysis Set (FAS)) | 77 (Number in Full Analysis Set (FAS))
Completed | 51 | 59
Not Completed | 24 | 18
Not completed — Adverse Event | 9 | 9
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 5 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lack of Efficacy | 6 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.4) | 35.9 (9.7) | 36.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 65 | 71 | 136
Log10 HIV viral load [Mean (Standard Deviation); unit: copies/mL] | 4.9 (0.8) | 4.9 (0.7) | 4.9 (0.8)
CD4+ count [Mean (Standard Deviation); unit: cells/mm^3] | 178.9 (105.3) | 183.5 (111.3) | 181.2 (108.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Response (VR)
Description: VR is defined as HIV viral load of <50 copies/ml measured at two consecutive visits PRIOR TO Week 48 and without subsequent rebound or change of ARV therapy prior to Week 48.
Time Frame: baseline to week 48
Population: All treated patients. Early withdrawals were considered failures.
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
participants
  Responders | 46 | 50
  Nonresponders | 29 | 27
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; With 75 evaluable patients per treatment group, this study had 80% power to observe a difference no lower than -6.5% assuming the true proportions of responders are both 65%; Test type: Non-Inferiority or Equivalence — A point estimate of -6.5% or higher for the diff. in the prop. of responders (NVP - ATV/r) was to be considered consistent with a successful ArTEN study. In the worst case for both studies, if the 2 studies were to be pooled, the non-inferiority margin of -12% would then be outside the 95% confidence interval (CI); p = 0.7142, Cochran-Mantel-Haenszel; Controlling for screening viral load and CD4+ categories; Difference in proportion of responders = -0.041, 95% CI [-0.183 to 0.101]

2. Secondary Outcome: Number of Participants With Virologic Response According to the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: HIV viral load <50 copies/ml measured at two consecutive visits UP TO Week 48 and without subsequent rebound or change of ARV therapy up to Week 48.
Time Frame: baseline to week 48
Population: All treated patients. Early withdrawals were considered failures.
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  Responders | 48 | 51
  Nonresponders | 27 | 26
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Non-Inferiority or Equivalence — Same as for the primary analysis; p = 0.6479, Cochran-Mantel-Haenszel; Controlling for screening viral load and CD4+ categories; Difference in proportion of responders = -0.027, 95% CI [-0.167 to 0.113]

3. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 48
Description: HIV viral load <50 copies/ml measured at Week 48 among observed cases on-treatment.
Time Frame: baseline to week 48
Population: Only includes treated patients with data in the Week 48 time window.
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  Responders | 42 | 48
  Nonresponders | 2 | 8
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Non-Inferiority or Equivalence — Same as for primary analysis; p = 0.1477, Cochran-Mantel-Haenszel; Controlling for screening viral load and CD4+ categories; Difference in proportion of responders = 0.084, 95% CI [-0.030 to 0.197]

4. Secondary Outcome: Number of Participants With Virologic Success (FDA Definition)
Description: HIV viral load <50 copies/ml measured in the Week 48 window whereby patients withdrawing early and patients without a Week 48 assessment are considered failures. Includes all participants in full analysis set (FAS).
Time Frame: baseline to week 48
Population: All treated patients.
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  Responders | 42 | 48
  Nonresponders | 33 | 29
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Non-Inferiority or Equivalence — Same as for primary analysis; p = 0.3703, Cochran-Mantel-Haenszel; Controlling for screening viral load and CD4+ categories; Difference in proportion of responders = -0.067, 95% CI [-0.215 to 0.080]

5. Secondary Outcome: Time to Virologic Response (First Confirmed Viral Load < 50 Copies/ml), All Participants
Description: Time to response whereby patients withdrawing early were censored after their withdrawal
Time Frame: baseline to week 48
Population: All treated patients
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
days | 57 [42 to 168] | 84 [56 to 173]
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Hazard ratio Atazanavir plus ritonavir / Nevirapine. Values < 1 indicate faster response in nevirapine; Test type: Superiority or Other; p = 0.0314, Regression, Cox; Controlling for screening viral load and CD4+ categories; Hazard Ratio (HR) = 0.666, 95% CI [0.460 to 0.964]

6. Secondary Outcome: Time to Virologic Response (First Confirmed Viral Load < 50 Copies/ml), Only Participants With Confirmed Viral Load < 50 Copies/ml
Time Frame: baseline to week 48
Population: All responders
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 55 | 65
days | 55 [41 to 85] | 84 [56 to 169]
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Responders only Hazard ratio Atazanavir plus ritonavir / Nevirapine. Values < 1 indicate faster response in nevirapine; Test type: Superiority or Other; p = 0.0172, Regression, Cox; Controlling for screening viral load and CD4+ categories; Hazard Ratio (HR) = 0.628, 95% CI [0.428 to 0.921]

7. Secondary Outcome: Number of Participants With Loss of Virologic Response Following Confirmed Virologic Response
Description: HIV viral load > 50 copies/ml on two consecutive measurements separated by at least 2 weeks, after confirmed virologic response (2 consecutive HIV viral load values < 50 copies/ml)
Time Frame: baseline to week 24 and week 48
Population: All treated patients; Too few patients had a loss of virologic response for a reasonable analysis of time to loss.
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  At week 24 | 1 | 4
  At week 48 | 2 | 9

8. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 2 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 2
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 6 | 5
  HIV viral load ≥ 50 copies/ml | 62 | 63
  Missing data | 7 | 9

9. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 4 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 4
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 12 | 10
  HIV viral load ≥ 50 copies/ml | 53 | 62
  Missing data | 10 | 5

10. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 6 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 6
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 23 | 14
  HIV viral load ≥ 50 copies/ml | 38 | 53
  Missing data | 14 | 10

11. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 8 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 8
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 34 | 23
  HIV viral load ≥ 50 copies/ml | 25 | 50
  Missing data | 16 | 4

12. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 12 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 12
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 42 | 43
  HIV viral load ≥ 50 copies/ml | 20 | 27
  Missing data | 13 | 7

13. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 24 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 24
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 48 | 61
  HIV viral load ≥ 50 copies/ml | 9 | 5
  Missing data | 18 | 11

14. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 36 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 36
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 53 | 55
  HIV viral load ≥ 50 copies/ml | 4 | 5
  Missing data | 18 | 17

15. Secondary Outcome: Number of Participants With HIV Viral Load < 50 Copies/ml at Week 48 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 48
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 50 copies/ml | 42 | 48
  HIV viral load ≥ 50 copies/ml | 2 | 8
  Missing data | 31 | 21

16. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 2 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 2
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 24 | 17
  HIV viral load ≥ 400 copies/ml | 44 | 51
  Missing data | 7 | 9

17. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 4 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 4
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 38 | 31
  HIV viral load ≥ 400 copies/ml | 27 | 41
  Missing data | 10 | 5

18. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 6 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 6
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 40 | 44
  HIV viral load ≥ 400 copies/ml | 21 | 23
  Missing data | 14 | 10

19. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 8 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 8
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 48 | 58
  HIV viral load ≥ 400 copies/ml | 11 | 15
  Missing data | 16 | 4

20. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 12 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 12
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 56 | 63
  HIV viral load ≥ 400 copies/ml | 6 | 7
  Missing data | 13 | 7

21. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 24 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 24
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 51 | 63
  HIV viral load ≥ 400 copies/ml | 6 | 3
  Missing data | 18 | 11

22. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 36 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 36
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 54 | 59
  HIV viral load ≥ 400 copies/ml | 3 | 1
  Missing data | 18 | 17

23. Secondary Outcome: Number of Participants With HIV Viral Load < 400 Copies/ml at Week 48 of Treatment
Description: Results within time windows, patients on-treatment
Time Frame: baseline to week 48
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  HIV viral load < 400 copies/ml | 43 | 54
  HIV viral load ≥ 400 copies/ml | 1 | 2
  Missing data | 31 | 21

24. Secondary Outcome: Number of Patients With Virologic Rebound to >400 Copies/ml
Description: HIV viral load >400 copies/ml on two consecutive measurements separated by at least 2 weeks, after confirmed virologic response (2 consecutive HIV viral load values < 50 copies/ml)
Time Frame: baseline to week 48
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants
  Rebound following response | 2 | 6
  No rebound following response | 55 | 63

25. Secondary Outcome: AIDS Progression and Death: Number of Patients With a Treatment-emergent AIDS Defining Illness or an AIDS-defining Illness Leading to Death
Description: AIDS defining illnesses include: Aspergillosis, Bartonellosis, Candidiasis, Cervical cancer, Chagas disease, Coccidiodomycosis, Cryptococcosis, Cytomegalovirus retinus, encephalopathy, Herpes Simplex Virus, Histoplasmosis, Isosporiasis, Kaposi's sarcoma, Leishmaniasis, Microsporidiosis, Mycobacterium avium complex, mycobacterium (non-tuberculous), Nocardiosis, Pneumocystis carinii pneumonia, Pneumonia, Progressive Multifocal Leukoencephalopathy, Rhodococcus equi, Salmonella, Toxoplasmosis, Wasting.
  Number of cases (no time-to analysis was performed due to small numbers).
Time Frame: baseline to week 48
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
Participants | 1 | 3

26. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 2.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 2
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 64 | 64
cells/mm^3 | 62.6 (80.9) | 61.0 (69.7)

27. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 4.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 4
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 65 | 70
cells/mm^3 | 76.4 (88.2) | 63.0 (72.6)

28. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 6.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 6
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 59 | 62
cells/mm^3 | 87.2 (86.0) | 78.4 (67.6)

29. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 8.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 8
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 58 | 69
cells/mm^3 | 111.9 (100.2) | 90.5 (85.2)

30. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 12.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 12
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 62 | 68
cells/mm^3 | 123.1 (109.5) | 102.2 (103.9)

31. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 24.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 24
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 59 | 68
cells/mm^3 | 131.8 (115.5) | 132.5 (86.8)

32. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 36.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 36
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 57 | 61
cells/mm^3 | 147.6 (120.7) | 120.5 (99.4)

33. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 48.
Description: Patients on-treatment, data within time windows
Time Frame: baseline to week 48
Population: Includes only treated patients with data in the specified time window
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 46 | 54
cells/mm^3 | 155.1 (118.8) | 160.4 (108.7)

34. Secondary Outcome: Change in Fasting Plasma Total Cholesterol Level
Time Frame: baseline to week 48
Population: All treated patients with data, Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 66 | 68
mg/dl | 18.2 (26.5) | 13.8 (39.5)
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Superiority or Other; p = 0.7315, ANCOVA; Controlling for screening viral load and CD4+ categories; Median Difference (Final Values) = 1.8, 95% CI [-8.4 to 11.9]

35. Secondary Outcome: Change in Fasting Plasma Triglycerides Level
Time Frame: baseline to week 48
Population: All treated patients with data, Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 66 | 68
mg/dl | -4.7 (87.6) | 8.4 (120.4)
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Superiority or Other; p = 0.3625, ANCOVA; Controlling for screening viral load and CD4+ categories; Median Difference (Final Values) = -10.6, 95% CI [-33.4 to 12.3]

36. Secondary Outcome: Change in Fasting High Density Lipoprotein (HDL) Cholesterol Level
Time Frame: baseline to week 48
Population: All treated patients with data, Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 66 | 68
mg/dl | 9.6 (11.8) | 3.5 (15.0)
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Superiority or Other; p = 0.0164, ANCOVA; Controlling for screening viral load and CD4+ categories; Mean Difference (Final Values) = 4.8, 95% CI [0.9 to 8.8]

37. Secondary Outcome: Change in Fasting Low Density Lipoprotein (LDL)Cholesterol Level
Time Frame: baseline to week 48
Population: All treated patients with data, Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 66 | 68
mg/dl | 8.7 (21.5) | 6.9 (32.2)
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Superiority or Other; p = 0.9257, ANCOVA; Controlling for screening viral load and CD4+ categories; Mean Difference (Final Values) = 0.4, 95% CI [-8.4 to 9.3]

38. Secondary Outcome: Change in Fasting Total Cholesterol to High Density Lipoprotein (HDL) Ratio
Time Frame: baseline to week 48
Population: All treated patients with data, Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 66 | 68
ratio | -0.38 (0.96) | -0.02 (1.06)
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Superiority or Other; p = 0.0375, ANCOVA; Controlling for screening viral load and CD4+ categories; Mean Difference (Final Values) = -0.33, 95% CI [-0.64 to -0.02]

39. Secondary Outcome: Change in Framingham Score
Description: Framingham prediction of 10-year risk of Coronary Heart Disease (CHD) outcomes (myocardial infarction [MI] or CHD death) based on the patient's gender, age, systolic blood pressure, total cholesterol, HDL-c and smoking status. The scale for the estimated risk ranges from 0 to 30%.
Time Frame: baseline to week 48
Population: All treated patients with data, Last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: percent 10-year risk
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 67 | 71
percent 10-year risk | -0.09 (2.01) | 0.14 (2.66)
Statistical Analysis 1: Comparison: Nevirapine (NVP) Plus Truvada vs Atazanavir Plus Ritonavir (ATV/r) Plus Truvada; Test type: Superiority or Other; p = 0.4645, ANCOVA; Controlling for screening viral load and CD4+ categories; Mean Difference (Final Values) = -0.28, 95% CI [-1.02 to 0.47]

40. Secondary Outcome: Change in Revised Framingham Score According to the Data Collection on Adverse Events of Anti-HIV Drugs (DAD) Study Group
Time Frame: baseline to week 48
Population: Not calculated as no data on family history of cardiovascular disease were available
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Change in Glomerular Filtration Rate (GFR) From Baseline to Week 48
Description: using 4-variable Modification of Diet in Renal Disease (MDRD) formula
Time Frame: baseline to week 48
Population: Includes only treated patients with data for the specified time window
Measure: Mean (Standard Deviation); unit: ml/min/1.73m^2
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 66 | 68
ml/min/1.73m^2 | -0.06 (33.90) | -12.81 (35.61)

42. Secondary Outcome: Percentage Adherence by Pill Count
Description: Number of pills not returned / number of treatment days in percent (%)
Time Frame: baseline to week 48
Population: All treated patients with data
Measure: Mean (Standard Deviation); unit: percentage adherence
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 71 | 76
percentage adherence | 94.3 (17.7) | 97.0 (8.1)

43. Secondary Outcome: Number of Participants With Genotypic Resistance at the Time of Virologic Failure.
Description: Genotypic resistance was measured by the following: Plasma samples for HIV-1 resistance were analyzed using a standard clinical assay that generates a virtual phenotypic interpretation of HIV-1 sequence data and predicts susceptibility or resistance of the isolate to approved ARVs. This analysis has not been performed.
Time Frame: baseline to week 48
Population: Includes only treated patients with data in the specified time window
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Incidence of Patients With AIDS Progression at Each Visit
Description: Cumulative incidence of patients with AIDS progression are shown
Time Frame: baseline to week 52
Population: Full Analysis set
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
participants
  week 0 | 0 | 0
  week 2 | 0 | 0
  week 4 | 0 | 0
  week 6 | 0 | 1
  week 8 | 0 | 1
  week 12 | 0 | 2
  week 24 | 0 | 3
  week 36 | 0 | 3
  week 48 | 1 | 3
  week 50 | 1 | 3
  End of Study Visit | 2 | 3

45. Secondary Outcome: Proportion of Patients Reporting CNS Side Effects of Any Severity
Time Frame: baseline to week 52
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
participants | 25 | 23

46. Secondary Outcome: Proportion of Patients Reporting Hepatic Events of Any Severity
Time Frame: baseline to week 52
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
participants | 5 | 24

47. Secondary Outcome: Proportion of Patients Reporting Rash of Any Severity
Time Frame: baseline to week 52
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
participants | 21 | 19

48. Secondary Outcome: Proportion of Patients With DAIDS Grade >= 2 Laboratory Abnormalities
Time Frame: baseline to week 52
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Number analyzed (Participants) | 75 | 77
participants
  Grade 2 moderate | 25 | 31
  Grade 3 severe | 8 | 7
  Grade 4 potential lifethreatening | 7 | 3

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Nevirapine (NVP) Plus Truvada | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada
Serious Adverse Events (participants affected / at risk) | 10/75 | 7/77
Other Adverse Events (participants affected / at risk) | 50/75 | 61/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine (NVP) Plus Truvada (N=75) | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada (N=77)
Bronchopneumonia (Infections and infestations) | 1 | 0
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Immune reconstitution syndrome (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Mononeuropathy multiplex (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nevirapine (NVP) Plus Truvada (N=75) | Atazanavir Plus Ritonavir (ATV/r) Plus Truvada (N=77)
Upper respiratory tract infection (Infections and infestations) | 8 | 18
Sinusitis (Infections and infestations) | 3 | 7
Anogenital warts (Infections and infestations) | 1 | 6
Bronchitis (Infections and infestations) | 2 | 5
Insomnia (Psychiatric disorders) | 4 | 7
Headache (Nervous system disorders) | 11 | 11
Dizziness (Nervous system disorders) | 4 | 5
Ocular icterus (Eye disorders) | 1 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 15
Nausea (Gastrointestinal disorders) | 10 | 11
Vomiting (Gastrointestinal disorders) | 3 | 6
Gastritis (Gastrointestinal disorders) | 0 | 4
Jaundice (Hepatobiliary disorders) | 0 | 12
Rash (Skin and subcutaneous tissue disorders) | 7 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Fatigue (General disorders) | 13 | 10
Oedema peripheral (General disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.